CLINICAL TRIAL: NCT03222921
Title: OpenGo Sensor Insole in Open Wedge HTO
Acronym: HTO
Status: Terminated | Type: Observational
Why Stopped: Technical issues, COVID-19
Sponsor: AO Innovation Translation Center (Other)
Collaborators: Berufsgenossenschaftlichen Unfallklinik Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: HTO Moticon
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2020-10

CONDITIONS: Tibia; Angulation
Keywords: high tibial osteotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: High tibial osteotomy — Patients undergoing high tibial osteotomy are investigated by a pressure insole for post-operative weight bearing behavior
  Other Names: pressure insole, OpenGo

SUMMARY:
Weight bearing in 40 patients undergoing open wedge high tibial osteotomy (HTO) will be studied during 12 weeks for their post-operative weight bearing using a pressure insole.

DETAILED DESCRIPTION:
Forty patients who are planned for open wedge HTO with deformity in the proximal tibia will be included in the study. The open wedge HTO will be performed in the well known biplanar technique and the TomoFix plate will be used as fixation plate. To analyze the peak pressure and if the patients are able to reassemble the partial weight bearing/ the full weight bearing the OpenGo Sensor Insole (Moticon) will be used during the first 12 weeks after surgery. In addition, x-rays will be analyze for the alignment and angles and clinical scores will be gathered to investigate patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Indication for high tibial osteotomy

Exclusion Criteria:

* Impairment of the shoulder which has an influence on the ability for partial weight bearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing high tibial osteotomy
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Partial weight bearing | 2 weeks post-OP
  Differences of the peak pressure (mean of the 13 pressure sensors) recorded by the insole vs. the recommended partial weight bearing of 20 kg and amount of events more than 20 kg partial weight bearing

SECONDARY OUTCOMES:
Full weight bearing | 12 weeks post-OP
  Time to full weight bearing after open wedge HTO
Weight bearing pre- vs. post-OP | 12 weeks post-OP
  Changes of peak pressure at the sole comparing varus deformity and after open wedge HTO
Patient reported outcomes | 12 weeks post-OP
  Depends the clinical outcome on the capability of early full-weight bearing?

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Simioni, Dr., Study Director — AO Clinical Investigation and Publishing Documentation
Locations (1):
- BGU Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided